CLINICAL TRIAL: NCT05802823
Title: The Effect of Standard Patient Simulation Method in Communication With Intensive Care Patients on Communication Skills, Satisfaction and Self-Confidence Levels in Learning of Nursing Students
Brief Title: Effects of Standard Patient Simulation Method in Communication With Intensive Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinop University (Other)
Responsible Party: Principal Investigator, Ümran Demircan, Lecturer, Sinop University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SINOPU
Record Dates: First submitted 2023-03-21; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Satisfaction; Communication; Confidence, Self
Keywords: simulated patient; communication; satisfaction
MeSH Terms: conditions — Personal Satisfaction; Communication

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Resources will be distributed to the students 1 week before the application, a scenario will be given 5 minutes before the application, and informed consent will be obtained from the students. Just before the application, information about the simulation process and analysis will be given. Students will be divided into 6 groups with the random numbers table and the application will be made on different days and times. The application time is 10-15 minutes and the camera will be recorded during the interview. At the end of the application, standard patient feedback will be given for each student. At the end of the application, analysis sessions will be held with the students as a group and feedback will be given by peers and trainers about their own performances. Analysis sessions will take between 30-45 minutes.
  Interventions: Other: Standardized Simülation Patient
- Control Group (No Intervention): No application will be made.

INTERVENTIONS:
Other: Standardized Simülation Patient — There are preliminary information, information, application and analysis sessions in the research. A rehearsal will be made 10 days before the application and arrangements will be made if necessary. The students will be given the resources 1 week before the application and the scenario 5 minutes before the application and informed consent will be obtained. Just before the application, information about the simulation process and analysis will be given. Students will be divided into 6 groups with the random numbers table and the application will be made on different days and times. The application time is 10-15 minutes and the camera will be recorded during the interview. At the end of the application, standard patient feedback will be given for each student. At the end of the application, analysis sessions will be held with the students as a group and feedback will be given by peers and trainers about their own performances. Analysis sessions will take between 30-45 minutes.
  Arms: Experimental Group

SUMMARY:
The research will be carried out in a randomized controlled experimental study design in order to evaluate the effect of standard patient simulation method on communication skills, satisfaction and self-confidence in learning of nursing students in communication with intensive care patients.

The research will be conducted face-to-face with nursing students who are in the 2nd year of the Faculty of Health Sciences of Sinop University and meet the inclusion criteria in the fall semester of 2022-2023, after the necessary permissions are obtained for the study.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of standard patient simulation method on communication skills, satisfaction and self-confidence in learning of nursing students in communication with intensive care patients.

Research hypotheses H0: The standard patient simulation method has no effect on the communication skills and satisfaction and self-confidence levels of nursing students in communication with intensive care patients.

H1: The standard patient simulation method has an effect on the communication skills and satisfaction and self-confidence levels of nursing students in communication with the intensive care patient.

Type of the study: The research will be carried out in a randomized controlled experimental study design in order to evaluate the effect of standard patient simulation method on communication skills, satisfaction and self-confidence in learning of nursing students in communication with intensive care patients.

Place and time of the research: The research will be conducted face-to-face with nursing students who are in the 2nd year of the Faculty of Health Sciences of Sinop University and meet the inclusion criteria in the fall semester of 2022-2023, after the necessary permissions are obtained for the study.

Population and Sample of the Research The universe of the research consists of one hundreds and three students who were studying in the second year of Sinop University Health Sciences Faculty Nursing Department and took the Communication Skills course in the fall semester of the 2022-2023 academic year. Power analysis in the study G Power 3.1.9.2. The sample size was calculated using the program. As a result of the analysis, it was determined that n=34 students in the intervention group and n=34 students in the control group should be included in the α=0.05 level, the effect size of 0.5 and 80% test power (Power 80%, alpha=0.05, effect size=0.5). In addition, considering the 10% possible losses in the implementation process, it was decided to have 38 people in each group. The study will be carried out with students who meet the inclusion criteria of the research among the students who make up the universe.

Data Collection Tools: The data of the study will be collected with the "Participant Information Form", "The Therapeutic Communication Skills Scale for Nursing Students" and "Student Satisfaction and Self Confidence in Learning Scale".

Introduction of Data Collection Tools

1. Participant Information Form: Participant information form prepared by the researcher; It includes the socio-demographic characteristics of University Students (age, gender, graduated school).
2. The Therapeutic Communication Skills Scale for Nursing Students (HÖTİBÖ): To measure students' therapeutic communication skills, is a seven-point Likert type (1=Never, 4=Sometimes 7=Always) that expresses how often the given proposition is used and consists of 16 questions. There are no reverse questions in the scale. HÖTİBÖ consists of three sub-dimensions: Nontherapeutic communication skills (seven items), Therapeutic communication skills-I (six items), Therapeutic communication skills-II (three items). Cronbach's alpha coefficient was calculated for the internal consistency reliability of the scale and the internal consistency coefficient of the 16-item scale was stated as .77. Internal consistency coefficient for each sub-dimension, Non-therapeutic communication skills .82; Therapeutic communication skills-I is .70 and Therapeutic communication skills-II is .60. A maximum of 112 and a minimum of 16 points can be obtained from the scale. As the score obtained from the sub-dimensions of the scale increases, it means that the students use the skills in that dimension more. In this study, the internal consistency coefficients are respectively; HÖTİBÖ 0.765, Non-therapeutic communication skills 0.753; Therapeutic communication skills-I were found to be 0.802 and Therapeutic communication skills-II were found to be 0.611. These values show that the Therapeutic Communication Skills Scale for Nursing Students is sufficient for the reliability level and gives stable results in each application of the scale.
3. Student Satisfaction and Self-Confidence in Learning Scale: The scale was developed by the National League for Nurses to measure students' attitudes and beliefs about simulation. The internal consistency coefficient of the scale, whose validity and reliability in Turkish was made by Karaçay and Kaya, was 0.88; 0.84 for student satisfaction sub-dimension and 0.83 for self-confidence in learning sub-dimension. The scale has two sub-dimensions: "satisfaction with learning" and "self-confidence". The total number of items is 13. In the sub-dimension of satisfaction with learning; Five items measuring satisfaction with the teaching method, variety of learning materials, facilitation, motivation, and the suitability of simulation in general, self-confidence sub-dimension; Content adequacy includes eight sub-items: self-confidence, content requirement, skill development, available resources, and information on how to get help to solve clinical problems in simulation. The 13th item in the scale was coded as reverse. The scale is answered as a five-point Likert (5= Strongly agree, 4=Agree, 3=Undecided: Neither agree nor disagree, 2=Disagree, 1=Strongly disagree). The score obtained is obtained from the sum of the items of the scale. A minimum score of 13 and a maximum score of 65 are obtained from the scale.

Application of Research This research will be carried out in two stages, namely preparation and implementation.

-Preparation Phase: Development of the Standard Patient Scenario: The application scenario will be prepared using the literature and based on the INACSL simulation application standards. The learning objectives of the Standard Patient simulation application are "Developing the ability of the student to initiate communication with the patient, identifying the factors that prevent / make it difficult to communicate with the patient in the intensive care unit, using non-verbal communication methods in his communication with the patient, predicting which therapeutic communication method to use according to the patient's reactions, nurse observation. and determining the nursing interventions according to the results of the evaluation, supporting the patient for cooperation in the implementation of the nursing interventions." determined as. The scenario design will be evaluated by field experts to cover the skills to achieve the learning objectives and necessary arrangements will be made. Scenario application visual sections are presented; It will consist of application steps in which student nurses are required to communicate with the intensive care patient in line with the correct procedure steps. Application link will be sent to students. The application time is fifteen minutes. The application scenario will be arranged in line with expert opinions.

Implementation Phase Pre-Test Application: Participant Information Form, Therapeutic Communication Skills Scale for Nursing Students will be pre-tested for all students in the study. Students to be included in the intervention and control groups will be assigned with the block randomization method according to the pre-test results. Students will not be informed which group they are in.

Standard Patient Simulation Practice: Standard patient method; Although it is a new and creative technique in which learning goals are determined, scenarios are created in which the characteristics of the patient and the patient's environment are presented, and standard patients belonging to the scenario are trained, students are recorded by interviewing standard patients in practice, and these recordings are monitored again and feedback is given. Thus, analysis sessions are held.

In the study, the students in the intervention group will participate in the preliminary information, prebriefing, application and debriefing sessions prepared by considering the scenario preparation criteria in the light of the literature.

Preparation of the Scenario: The simulation scenario and its contents will be prepared by experts in the field of psychiatric nursing, including the skills to achieve the determined learning objectives. The case scenarios to be used in standard patient practice were chosen to measure the skills they had difficulty with as a result of the feedback of the students who had practiced in previous years and the observations of the instructors. Actors trained to play the standard patient role will be used. The prepared case scenario will be given to the person playing the role of the standard patient 10 days before the application, and the content and flow of the scenario, the student group, the expected goals from the students, giving feedback and the things to be considered while animating the scenario will be discussed. Before the day of the practice of the study, a rehearsal will be held with the actor playing the role of the standard patient. In practice, the standard patient will be recorded with a volunteer student, feedback will be given to the standard patient through the recorded videos, and if necessary, re-arrangements will be made.

* Preliminary Preparation: Regarding the application process, the date, place, time and duration of the application will be explained to the students in a meeting by the researcher. Resources will be given to students 1 week before the application. Standard Patient method will be introduced.
* Prebriefing: Students will be given a scenario 5 minutes before the application and informed consent will be obtained from the students.
* Briefing: In order to standardize the education method given to the students, a meeting will be held by the researcher just before the application, where information about the place and time of the simulation process and the analysis interviews to be held after the application, and the students' questions will be answered.
* Making the Application: In accordance with the number of students, the students will be divided into 6 groups using a random number table, in accordance with the standards determined by the INACSL Standards Committee, in a way that prevents the communication of students with each other. The application will be made on different days and times. 10-15 minutes will be allocated for each student's interview, and recording will be made with the help of a camera during the interview. At the end of the simulation, the standard patient will give feedback on the performance of each of the students.
* Debriefing: After the application is completed, debriefing sessions will be held with the students as a group and feedback will be given by peers and trainers about their own performances. Feedback will be non-judgmental and positive. Students will be asked for their opinions about their experiences in the analysis session. Analysis sessions will be held between 30-45 minutes in the light of the application criteria in the literature.

Post-Test Application: Post-Test Application In line with the opinions of the experts in the field of Biostatistics and Measurement and Evaluation, two weeks after the simulation application, the Therapeutic Communication Skills Scale for Nursing Students, Student Satisfaction and Self-Confidence in Learning Scale will be administered to the students in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

Having taken the course of Self-Knowledge and Communication Methods, Those who have not participated in a practical activity (course, simulation application, applied program, etc.) for communication skills No experience working in the intensive care unit 18 years and over, No written or verbal communication problems, Students who volunteer to participate in the research will be included in the research.

Exclusion Criteria:

* Having a psychiatric or neurological disease that will prevent the understanding and interpretation of the simulation application, Students who have problems in speaking/understanding Turkish will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-04-25 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Communication Evaluated Using The Therapeutic Communication Skills Scale for Nursing Students | change from before implication and 3 th week of practice
  Scores ranging from 16 to 112 points are obtained in the scale.

SECONDARY OUTCOMES:
Nurses to measure students' attitudes and beliefs about simulation using Student Satisfaction and Self-Confidence in Learning Scale | change from before implication and 3 th week of practice
  Scores ranging from 13 to 65 points are obtained in the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF